CLINICAL TRIAL: NCT04451707
Title: Multicentre Retrospective Study on the Clinical and Epidemiological Characteristics and Therapeutic Management of Non-cholera Vibrio Infections
Brief Title: Epidemiology Non-cholera Vibrio Infections
Acronym: INFECTIVE
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/P02/358
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Vibrio Infections
MeSH Terms: conditions — Vibrio Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-cholera Vibrio infection: Patients diagnosed with non-cholera Vibrio infection in Western France from 2000 to 2019
  Interventions: Other: non-cholera Vibrio infection

INTERVENTIONS:
Other: non-cholera Vibrio infection — Epidemiology of patients diagnosed with non-cholera Vibrio infection

SUMMARY:
The purpose of this study is to identify the epidemiological and clinical characteristics of patients diagnosed with non-cholera Vibrio infection in Western France from 2000 to 2019.

DETAILED DESCRIPTION:
Vibrios are gram-negative, ubiquitous bacteria of the marine flora and are found particularly in warm waters. For example, the incidence is high in Florida and Vibrio infections are now reportable in the United States. Different species of Vibrio are described. A distinction is made between choleric vibrios belonging to serogroups O1 and O139, responsible for cholera epidemics, and non-choleric vibrios. Our study will focus on non-cholera vibrios. Vibrio infections can occur by eating contaminated raw seafood or by exposure of a wound to the marine environment. They occur mainly during the hot summer months. This can be explained on the one hand by higher water temperature and on the other hand by increased beach use. With global warming, it is possible that Vibrio infections may increase in number and location.

ELIGIBILITY:
Inclusion Criteria:

* non-cholera Vibrio infection

Exclusion Criteria:

* vibriosis to Vibrio cholerae O1 and O139

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-cholera Vibrio infection in Western France from 2000 to 2019
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Hoefler, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (7):
- France (7):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - Centre Hospitalier Départemental de la Vendée, La Roche-sur-Yon
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available with publication. Keyword are infection, non-cholera Vibrio, epidemiology The only available version will be the locked database. The database will be made available by the study director upon request up to 15 years after publication.
  Medical Subject Headings (MESH) terms will be used to describe clinical data. Methodology for will be provided in the publication. International standard unit will be used.
Supporting Information: CSR
Time Frame: From publication and up to 15 years after publication
Access Criteria: Contact the corresponding author of the publication

REFERENCES:
- [Background] Weis KE, Hammond RM, Hutchinson R, Blackmore CG. Vibrio illness in Florida, 1998-2007. Epidemiol Infect. 2011 Apr;139(4):591-8. doi: 10.1017/S0950268810001354. Epub 2010 Jun 14. PMID 20546636
- [Background] Morris JG Jr. Cholera and other types of vibriosis: a story of human pandemics and oysters on the half shell. Clin Infect Dis. 2003 Jul 15;37(2):272-80. doi: 10.1086/375600. Epub 2003 Jul 3. PMID 12856219
- [Background] Givens CE, Bowers JC, DePaola A, Hollibaugh JT, Jones JL. Occurrence and distribution of Vibrio vulnificus and Vibrio parahaemolyticus--potential roles for fish, oyster, sediment and water. Lett Appl Microbiol. 2014 Jun;58(6):503-10. doi: 10.1111/lam.12226. Epub 2014 Feb 27. PMID 24571291
- [Background] Jones MK, Oliver JD. Vibrio vulnificus: disease and pathogenesis. Infect Immun. 2009 May;77(5):1723-33. doi: 10.1128/IAI.01046-08. Epub 2009 Mar 2. No abstract available. PMID 19255188
- [Result] Hoefler F, Pouget-Abadie X, Roncato-Saberan M, Lemarie R, Takoudju EM, Raffi F, Corvec S, Le Bras M, Cazanave C, Lehours P, Guimard T, Allix-Beguec C. Clinical and Epidemiologic Characteristics and Therapeutic Management of Patients with Vibrio Infections, Bay of Biscay, France, 2001-2019. Emerg Infect Dis. 2022 Dec;28(12):2367-73. doi: 10.3201/eid2812.220748. PMID 36418019

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-cholerae or Non-O1/O139 Vibrio Infection: Epidemiology of patients diagnosed with non-cholerae or non-O1/O139 Vibrio infection in Western France from 2000 to 2019
Period: Overall Study
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
Started | 67
Completed | 67
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Non-cholera Vibrio Infection
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 28
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (24.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 67
Region of Enrollment [Number; unit: participants]
  France | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Diagnosed Non-cholerae or Non-O1/O139 Vibrio Infection
Description: A non-cholerae or non-O1/O139 Vibrio infection was defined by a biological sample (blood, superficial sample, deep sample, and ear sample) positive to a Vibrio species other than Vibrio cholerae O1-O139.
Time Frame: Up to 20 years, from 2000-2019
Measure: Count of Participants; unit: Participants
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
Number analyzed (Participants) | 67
Participants
  Center 1 | 20
  Center 2 | 7
  Center 3 | 2
  Center 4 | 18
  Center 5 | 10
  Center 6 | 1
  Center 7 | 1
  Center 8 | 8

2. Secondary Outcome: Number of Patients Per Clinical History
Description: Clinical history: diabetes, heart failure, hepatopathy, neoplasia, alcohol use disorder, Immunosuppressive drug, Pre-existing wound, Digestive surgery, Hemopathy, Kidney Disease
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
Number analyzed (Participants) | 67
Participants
  Heart failure | 24
  Neoplasia | 11
  Diabetes | 8
  kidney failure | 7
  Immune disease | 7
  Haemopathy | 5
  Liver disease | 5
  Alcohol use disorder | 7
  Pre-existing wound | 6
  Digestive surgery | 6

3. Secondary Outcome: Number of Participants Associated With Environmental Factors
Description: environmental factors : seafood consumption, bathing/water activity, Injury in the aquatic environment, Walk to the beach, Handling of seafood products, returning from a trip abroad
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
Number analyzed (Participants) | 67
Participants
  Bathing in the sea | 12
  Injury in the aquatic environment | 5
  Aquatic activities | 3
  Walk on the beach | 2
  Seafood consumption | 7
  Handling of seafood products | 7
  Returning from a trip abroad | 2
  Unknown | 29

4. Secondary Outcome: Number of Participants Per Identified Species
Description: Species: Vibrio alginolyticus, Vibrio cholerae Non-O1/Non-O139 Non toxinogenic, Vibrio parahaemolyticus, Vibrio vulnificus, Vibrio sp or other
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
Number analyzed (Participants) | 67
Participants
  Vibrio alginolyticus | 23
  Vibrio parahaemolyticus | 20
  Non-O1/O139 Vibrio cholerae | 10
  Vibrio vulnificus | 7
  Vibrio spp | 7

5. Secondary Outcome: Number of Participants by Month of the Years
Time Frame: at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
Number analyzed (Participants) | 67
Participants
  January | 0
  February | 0
  March | 1
  April | 0
  May | 1
  June | 6
  July | 14
  August | 19
  September | 11
  October | 6
  Novermber | 2
  December | 1
  Unknown | 6

6. Secondary Outcome: Number of Participants Treated by Antibiotics
Time Frame: through study completion, an average of 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
Number analyzed (Participants) | 67
Participants
  Treated by antibiotics | 53
  Did not received antibiotics | 5
  unknown | 9

7. Secondary Outcome: Number of Participants Per Outcome
Description: outcome :cure, cure with amputation, and deceased due to the infection
Time Frame: through study completion, an average of 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
Number analyzed (Participants) | 67
Participants
  Cured | 53
  Amputation | 6
  Infection related death | 8

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | Non-cholerae or Non-O1/O139 Vibrio Infection
All-Cause Mortality (participants affected / at risk) | 8/67
Serious Adverse Events (participants affected / at risk) | 35/67
Other Adverse Events (participants affected / at risk) | 41/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-cholerae or Non-O1/O139 Vibrio Infection (N=67)
Amputation (Infections and infestations) | 6
Surgery (Infections and infestations) | 21
Near Drowning (Infections and infestations) | 3
Abdominal and gastrointestinal infection (Infections and infestations) | 1 — Severe infection in a patient with cancer
Septic shock (Infections and infestations) | 3
Necrotizing fasciitis (Infections and infestations) | 1 — patient with blood disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-cholerae or Non-O1/O139 Vibrio Infection (N=67)
Fever (Infections and infestations) | 29
Abdominal crampy pain (Infections and infestations) | 20
Diarrhea (Infections and infestations) | 19
Vomiting (Infections and infestations) | 13
Nausea (Infections and infestations) | 11
Headache (Infections and infestations) | 2
Dyspnea (Infections and infestations) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT04451707/Prot_SAP_000.pdf